CLINICAL TRIAL: NCT04349072
Title: A Randomized, Double-blind, Placebo-controlled Study to Evaluate Mavacamten in Adults With Symptomatic Obstructive Hypertrophic Cardiomyopathy Who Are Eligible for Septal Reduction Therapy
Brief Title: A Study to Evaluate Mavacamten in Adults With Symptomatic Obstructive HCM Who Are Eligible for Septal Reduction Therapy
Acronym: VALOR-HCM
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CV027-006
Record Dates: First submitted 2020-04-07; First posted 2020-04-16 (Actual); Results first posted 2023-03-07 (Actual); Last update posted 2025-05-23 (Actual); Status verified 2025-05

CONDITIONS: HOCM, Hypertrophic Obstructive Cardiomyopathy
MeSH Terms: conditions — Cardiomyopathy, Hypertrophic | interventions — MYK-461

STUDY DESIGN:
Intervention Model Description: This is a parallel group treatment study with 2 treatment groups; subjects and investigators are blinded to treatment and dose for the first 16 weeks of treatment. Mavacamten dose is blinded throughout the study.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Drug: Mavacamten (Experimental): Mavacamten Capsules
  Other names:
  MYK-461
  Interventions: Drug: Mavacamten
- Drug: Placebo (Placebo Comparator): Matching Placebo Capsules
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Mavacamten — Mavacamten Capsules Other names: MYK-461
  Arms: Drug: Mavacamten
Drug: Placebo — Placebo
  Arms: Drug: Placebo

SUMMARY:
This is a randomized, double-blind, placebo-controlled, multi-center study in the United States (U.S.) that will evaluate the effect of mavacamten treatment on reducing the number of septal reduction therapy (SRT) procedures performed in subjects with symptomatic obstructive hypertrophic cardiomyopathy (oHCM [also known as HOCM]) who are eligible for SRT based on ACCF/AHA 2011 and/or ESC 2014 guidelines.

ELIGIBILITY:
Key Inclusion Criteria:

* At least 18 years old at screening and body weight > 45 kg at screening
* Diagnosed with oHCM consistent with current ACCF/AHA 2011 and meet their recommendations for invasive therapies
* Referred or under active consideration within the past 12 months for SRT procedure and willing to have SRT procedure
* Has documented left ventricular ejection fraction (LVEF) ≥ 60% at Screening
* Has documented oxygen saturation at rest ≥ 90% at Screening

Key Exclusion Criteria:

* Persistent or permanent atrial fibrillation and subject not on anticoagulation for ≥ 4 weeks prior to screening and/or not adequately rate controlled ≤ 6 months prior to screening
* Previously treated with invasive septal reduction (surgical myectomy or percutaneous alcohol septal ablation [ASA])
* For individuals on beta blockers, calcium channel blockers, or disopyramide, any dose adjustment of these medications < 14 days prior to screening or an anticipated change in regimen during the first 16 weeks of the study
* Any medical condition that precludes upright exercise stress testing
* Paroxysmal, intermittent atrial fibrillation with atrial fibrillation present at screening
* Prior treatment with cardiotoxic agents, such as doxorubicin or similar
* Has a history or evidence of any other clinically significant disorder, condition, or disease that would pose a risk to subject safety or interfere with the study evaluation, procedures, or completion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 112 (Actual)
Dates: Start 2020-07-06 (Actual); Primary Completion 2022-02-07 (Actual); Study Completion 2024-05-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (21):
- United States (21):
  - Local Institution - 0009, Los Angeles, California
  - Local Institution - 0011, Stanford, California
  - Local Institution - 0001, New Haven, Connecticut
  - Local Institution - 0021, Weston, Florida
  - Local Institution - 0016, Boston, Massachusetts
  - Local Institution - 0007, Boston, Massachusetts
  - Local Institution - 0006, Ann Arbor, Michigan
  - Local Institution - 0013, Grand Rapids, Michigan
  - Local Institution - 0015, Rochester, Minnesota
  - Local Institution - 0005, St Louis, Missouri
  - Local Institution - 0010, New York, New York
  - Local Institution - 0017, Valhalla, New York
  - Local Institution - 0004, Durham, North Carolina
  - Local Institution - 0020, Cleveland, Ohio
  - Local Institution - 0002, Portland, Oregon
  - Local Institution - 0003, Philadelphia, Pennsylvania
  - Local Institution - 0019, Pittsburgh, Pennsylvania
  - Local Institution - 0014, Nashville, Tennessee
  - Local Institution - 0018, Nashville, Tennessee
  - Local Institution, Houston, Texas
  - Local Institution - 0012, Murray, Utah

REFERENCES:
- [Derived] Desai MY, Wolski K, Owens A, Geske JB, Saberi S, Wang A, Sherrid M, Cremer PC, Lakdawala NK, Tower-Rader A, Fermin D, Naidu SS, Smedira NG, Schaff H, Gong Z, Mudarris L, Lampl K, Sehnert AJ, Nissen SE; VALOR-HCM Investigators. Mavacamten in Patients With Hypertrophic Cardiomyopathy Referred for Septal Reduction: Week 128 Results From VALOR-HCM. Circulation. 2025 May 13;151(19):1378-1390. doi: 10.1161/CIRCULATIONAHA.124.072445. Epub 2024 Nov 18. PMID 39556124
- [Derived] Desai MY, Okushi Y, Wolski K, Geske JB, Owens A, Saberi S, Wang A, Cremer PC, Sherrid M, Lakdawala NK, Tower-Rader A, Fermin D, Naidu SS, Lampl KL, Sehnert AJ, Nissen SE, Popovic ZB; VALOR-HCM Investigators. Mavacamten-Associated Temporal Changes in Left Atrial Function in Obstructive HCM: Insights From the VALOR-HCM Trial. JACC Cardiovasc Imaging. 2025 Mar;18(3):251-262. doi: 10.1016/j.jcmg.2024.08.005. Epub 2024 Sep 2. PMID 39254622
- [Derived] Desai MY, Okushi Y, Gaballa A, Wang Q, Geske JB, Owens AT, Saberi S, Wang A, Cremer PC, Sherrid M, Lakdawala NK, Tower-Rader A, Fermin D, Naidu SS, Lampl KL, Sehnert AJ, Nissen SE, Popovic ZB; VALOR-HCM Investigators. Serial Changes in Ventricular Strain in Symptomatic Obstructive Hypertrophic Cardiomyopathy Treated With Mavacamten: Insights From the VALOR-HCM Trial. Circ Cardiovasc Imaging. 2024 Sep;17(9):e017185. doi: 10.1161/CIRCIMAGING.124.017185. Epub 2024 Sep 2. PMID 39221824
- [Derived] Desai MY, Owens A, Wolski K, Geske JB, Saberi S, Wang A, Sherrid M, Cremer PC, Lakdawala NK, Tower-Rader A, Fermin D, Naidu SS, Smedira NG, Schaff H, McErlean E, Sewell C, Mudarris L, Gong Z, Lampl K, Sehnert AJ, Nissen SE. Mavacamten in Patients With Hypertrophic Cardiomyopathy Referred for Septal Reduction: Week 56 Results From the VALOR-HCM Randomized Clinical Trial. JAMA Cardiol. 2023 Oct 1;8(10):968-977. doi: 10.1001/jamacardio.2023.3342. PMID 37639243
- [Derived] Cremer PC, Geske JB, Owens A, Jaber WA, Harb SC, Saberi S, Wang A, Sherrid M, Naidu SS, Schaff H, Smedira NG, Wang Q, Wolski K, Lampl KL, Sehnert AJ, Nissen SE, Desai MY. Myosin Inhibition and Left Ventricular Diastolic Function in Patients With Obstructive Hypertrophic Cardiomyopathy Referred for Septal Reduction Therapy: Insights From the VALOR-HCM Study. Circ Cardiovasc Imaging. 2022 Dec;15(12):e014986. doi: 10.1161/CIRCIMAGING.122.014986. Epub 2022 Nov 6. PMID 36335645
- [Derived] Desai MY, Owens A, Geske JB, Wolski K, Saberi S, Wang A, Sherrid M, Cremer PC, Naidu SS, Smedira NG, Schaff H, McErlean E, Sewell C, Balasubramanyam A, Lampl K, Sehnert AJ, Nissen SE. Dose-Blinded Myosin Inhibition in Patients With Obstructive Hypertrophic Cardiomyopathy Referred for Septal Reduction Therapy: Outcomes Through 32 Weeks. Circulation. 2023 Mar 14;147(11):850-863. doi: 10.1161/CIRCULATIONAHA.122.062534. Epub 2022 Nov 6. PMID 36335531
- [Derived] Desai MY, Owens A, Geske JB, Wolski K, Naidu SS, Smedira NG, Cremer PC, Schaff H, McErlean E, Sewell C, Li W, Sterling L, Lampl K, Edelberg JM, Sehnert AJ, Nissen SE. Myosin Inhibition in Patients With Obstructive Hypertrophic Cardiomyopathy Referred for Septal Reduction Therapy. J Am Coll Cardiol. 2022 Jul 12;80(2):95-108. doi: 10.1016/j.jacc.2022.04.048. PMID 35798455
- [Derived] Zampieri M, Argiro A, Marchi A, Berteotti M, Targetti M, Fornaro A, Tomberli A, Stefano P, Marchionni N, Olivotto I. Mavacamten, a Novel Therapeutic Strategy for Obstructive Hypertrophic Cardiomyopathy. Curr Cardiol Rep. 2021 Jun 3;23(7):79. doi: 10.1007/s11886-021-01508-0. PMID 34081217
- [Derived] Desai MY, Wolski K, Owens A, Naidu SS, Geske JB, Smedira NG, Schaff H, Lampl K, McErlean E, Sewell C, Zhang D, Edelberg JM, Sehnert AJ, Nissen SE. Study design and rationale of VALOR-HCM: evaluation of mavacamten in adults with symptomatic obstructive hypertrophic cardiomyopathy who are eligible for septal reduction therapy. Am Heart J. 2021 Sep;239:80-89. doi: 10.1016/j.ahj.2021.05.007. Epub 2021 May 24. PMID 34038706
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — http://www.BMSClinicalTrials.com

RESULTS

PARTICIPANT FLOW:
Groups:
- Mavacamten: Participants randomized to the mavacamten group started on 5 mg once daily and were titrated to receive 2.5, 5, 10, or 15 mg capsule orally once daily based on possible down-titration at Week 4 and up-titration at Weeks 8 and 12 (based on the LVEF and VLVOT gradient measured by TTE). Participants could be up- titrated at any scheduled visit after Week 32.
  Participants went through 16 weeks of placebo-controlled treatment (Day 1 to Week 16), 16 weeks of active-controlled treatment (Weeks 16 to 32), and 96 weeks of LTE mavacamten (Weeks 32 to 128).
- Placebo to Mavacamten: One placebo-to-match mavacamten capsule once daily for 16 weeks and then switch to mavacamten. After Week 16 through Week 32, participants started on 5 mg once daily and were titrated to receive 2.5, 5, 10, or 15 mg capsule orally once daily based on possible down-titration at Week 20 and up-titration at Weeks 24 and 28 (based on the LVEF and VLVOT gradient measured by TTE). Participants could be up- titrated at any scheduled visit after Week 32.
  Participants went through 16 weeks of placebo-controlled treatment (Day 1 to Week 16), 16 weeks of active-controlled treatment (Weeks 16 to 32), and 96 weeks of LTE mavacamten (Weeks 32 to 128).
Period: Randomization Period
Arm/Group | Mavacamten | Placebo to Mavacamten
Started | 56 | 56
Completed | 56 | 55
Not Completed | 0 | 1
Period: Double Blind Treatment Period
Arm/Group | Mavacamten | Placebo to Mavacamten
Started | 56 | 55
Completed (Ongoing treatment) | 52 | 45
Not Completed | 4 | 10
Period: Long Term Follow up
Arm/Group | Mavacamten | Placebo to Mavacamten
Started | 56 | 52
Completed | 51 | 42
Not Completed | 5 | 10

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Mavacamten | Placebo to Mavacamten | Total
Number analyzed (Participants) | 56 | 56 | 112
Age, Continuous [Mean (Standard Deviation); unit: Years] | 59.8 (14.18) | 60.9 (10.55) | 60.3 (12.45)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27 | 28 | 55
  Male | 29 | 28 | 57
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1
  Not Hispanic or Latino | 56 | 54 | 110
  Unknown or Not Reported | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 2 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 0 | 3
  White | 48 | 52 | 100
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 3 | 3 | 6

OUTCOME MEASURES:

1. Primary Outcome: Composite of Decision to Proceed With Septal Reduction Therapy (SRT) and SRT Guideline Eligible at Week 16
Description: Participants who decided to proceed with SRT or were eligible for SRT at week 16. Participants with missing assessments were classified as meeting the primary endpoint (did not improve).
  SRT eligibility using the New York Heart Association Functional Class (NYHA) and left ventricular outflow tract (LVOT) assessments per the 2011 ACCF/AHA guideline clinical and hemodynamic criterion are below:
  * NYHA Class III or IV/ NYHA Class II with exertion-induced syncope/near syncope, AND
  * Dynamic LVOT gradient at rest or with provocation >= 50 mmHg.
  NYHA Class II at week 16, the following rules will be applied:
  * NYHA Class II with history of exertional syncope/ syncope at baseline and at W16 is still NYHA Class II, they remain SRT eligible IF their maximal LVOT gradient is ≥ 50mmHg
  * NYHA Class III/IV at baseline and at W16 has improved to Class II, they are no longer SRT eligible UNLESS they have AE of exertional syncope or pre-syncope during the 16 weeks.
Time Frame: Week 16
Population: All randomized participants
Measure: Count of Participants; unit: Participants
Arm/Group | Mavacamten | Placebo to Mavacamten
Number analyzed (Participants) | 56 | 56
Participants | 10 | 43
Statistical Analysis 1: Comparison: Mavacamten vs Placebo to Mavacamten; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel; Proportion Difference = 58.93, 95% CI 2-sided [43.989 to 73.868]

2. Secondary Outcome: Number of Participants With at Least One Class Improvement From Baseline in New York Heart Association (NYHA) Class at Week 16
Description: The NYHA functional classification of heart failure assigns participants to 1 of 4 categories based on the participants symptoms. Baseline values are defined generally as the last available value before the first administration of study drug of analysis interest. Participants with missing NYHA class assessments are treated as no improvement.
  Class 1: No limitation of physical activity. Ordinary physical activity does not cause undue fatigue, palpitation, dyspnea (shortness of breath).
  Class 2: Slight limitation of physical activity. Comfortable at rest. Ordinary physical activity results in fatigue, palpitation, dyspnea (shortness of breath).
  Class 3: Marked limitation of physical activity. Comfortable at rest. Less-than ordinary-activity causes fatigue, palpitation, or dyspnea. Class 4: Unable to carry on any physical activity without discomfort. Symptoms of heart failure at rest. If any physical activity is undertaken, discomfort increases.
Time Frame: Baseline and week 16
Population: All randomized participants
Measure: Count of Participants; unit: Participants
Arm/Group | Mavacamten | Placebo to Mavacamten
Number analyzed (Participants) | 56 | 56
Participants | 35 | 12
Statistical Analysis 1: Comparison: Mavacamten vs Placebo to Mavacamten; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel; Proportion Difference = 41.07, 95% CI 2-sided [24.481 to 57.662]

3. Secondary Outcome: Change From Baseline to Week 16 in Kansas City Cardiomyopathy Questionnaire 23-item Version, Clinical Summary Score (KCCQ-23, CSS)
Description: The KCCQ-23 is a 23-item, self-administered questionnaire that measures the impact of a participant's cardiovascular disease or its treatment on 6 distinct domains using a 2-week recall period: symptoms/signs, physical limitation, quality of life (QoL), social limitations, self-efficacy, and symptom stability. The KCCQ 23 Clinical Summary Score (CSS) is derived from the Total Symptom Score (TSS) and the Physical Limitations (PL) score of the KCCQ 23. The CSS, TSS, and the PL score range from 0 to 100 with higher scores representing less severe symptoms and/or physical limitations. The CSS is a mean of the TSS and the PL score.
Time Frame: Baseline and week 16
Population: All randomized participants with baseline and week 16 clinical summary scores
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Mavacamten | Placebo to Mavacamten
Number analyzed (Participants) | 55 | 53
Score on a scale | 10.4 (16.06) | 1.8 (12.01)
Statistical Analysis 1: Comparison: Mavacamten vs Placebo to Mavacamten; Test type: Superiority; p < 0.0001, Mixed Models Analysis; Mixed model with repeated measure (MMRM); Leat Square Mean of Treatment Difference = 9.45, 95% CI 2-sided [4.868 to 14.041]

4. Secondary Outcome: Change From Baseline to Week 16 in N-Terminal Pro-b-Type Natriuretic Peptide (NT-proBNP)
Description: A geometric mean ratio was used to assess the change from baseline to Week 16 in N-Terminal Pro-b-Type Natriuretic Peptide (NT-proBNP). Baseline values are defined as the last non-missing value prior to the first dose of study drug unless specified otherwise.
Time Frame: Baseline and week 16
Population: All randomized participants with baseline and week 16 serum concentration data
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/L
Arm/Group | Mavacamten | Placebo to Mavacamten
Number analyzed (Participants) | 55 | 53
ng/L | 0.35 (NA) — Geometric coefficient of variation was not calculated and the arithmetic coefficient of variation (% CV) is being reported. %CV = 83.677 | 1.13 (NA) — Geometric coefficient of variation was not calculated and the arithmetic coefficient of variation (% CV) is being reported. %CV = 57.809
Statistical Analysis 1: Comparison: Mavacamten vs Placebo to Mavacamten; Test type: Superiority; p < 0.0001, Mixed Models Analysis; Mixed model with repeated measure (MMRM); Mean Ratio = 0.33, 95% CI 2-sided [0.266 to 0.421]

5. Secondary Outcome: Change From Baseline to Week 16 in Cardiac Troponin
Description: A geometric mean ratio was used to assess the change from baseline to week 16 in cardiac troponin. Baseline values are defined as the last non-missing value prior to the first dose of study drug unless specified otherwise.
Time Frame: Baseline and week 16
Population: All randomized participants with baseline and week 16 serum concentration data
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/L
Arm/Group | Mavacamten | Placebo to Mavacamten
Number analyzed (Participants) | 55 | 53
ng/L | 0.50 (NA) — Geometric coefficient of variation was not calculated and the arithmetic coefficient of variation (% CV) is being reported. %CV = 100.992 | 1.03 (NA) — Geometric coefficient of variation was not calculated and the arithmetic coefficient of variation (% CV) is being reported. %CV = 85.716
Statistical Analysis 1: Comparison: Mavacamten vs Placebo to Mavacamten; Test type: Superiority; p < 0.0001, Mixed Models Analysis; Mixed model with repeated measure (MMRM); Mean Ratio = 0.53, 95% CI 2-sided [0.406 to 0.700]

6. Secondary Outcome: Change From Baseline to Week 16 in Post-Exercise Left Ventricular Outflow Tract (LVOT) Gradient
Description: Change from baseline to week 16 in post-exercise left ventricular outflow tract (LVOT) gradient. Baseline values are defined as the last non-missing value prior to the first dose of study drug unless specified otherwise.
Time Frame: Baseline and week 16
Population: All randomized participants with baseline and week 16 measurements
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Mavacamten | Placebo to Mavacamten
Number analyzed (Participants) | 55 | 53
mmHg | -39.1 (36.51) | -1.8 (28.82)
Statistical Analysis 1: Comparison: Mavacamten vs Placebo to Mavacamten; Test type: Superiority; p < 0.0001, ANCOVA; Leat Square Mean of Treatment Difference = -37.2, 95% CI 2-sided [-48.08 to -26.24]

ADVERSE EVENTS:
Time Frame: Other (Not including Serious) Adverse Events (AEs) and Serious Adverse Events (SAEs) are collected from first dose to 56 days post last dose (Up to approximately 146 weeks). Participants were assessed for All-cause mortality from their date of randomization to study completion (Up to approximately 46 months.)
Description: The number at Risk for All-Cause Mortality represents all Randomized Participants. The number at Risk for Serious Adverse Events and Other (Not Including Serious) Adverse Events represents all participants that received at least 1 dose of study medication.
  108 participants in total received mavacamtem (56 participants who started treatment with mavacamten plus the 52 participants who originally received placebo and switched over at week 16).
Groups:
- Mavacamten: Participants started on 5 mg once daily and were titrated to receive 2.5, 5, 10, or 15 mg capsule orally once daily based on possible down-titration and up-titration (based on the LVEF and VLVOT gradient measured by TTE).
- Placebo: One placebo-to-match mavacamten capsule once daily for 16 weeks.
Arm/Group | Mavacamten | Placebo
All-Cause Mortality (participants affected / at risk) | 1/108 | 0/56
Serious Adverse Events (participants affected / at risk) | 21/108 | 1/55
Other Adverse Events (participants affected / at risk) | 96/108 | 20/55
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Mavacamten (N=108) | Placebo (N=55)
Acute left ventricular failure (Cardiac disorders) | 1 | 0
Acute myocardial infarction (Cardiac disorders) | 1 | 0
Arrhythmia (Cardiac disorders) | 1 | 0
Atrial fibrillation (Cardiac disorders) | 4 | 0
Bradycardia (Cardiac disorders) | 1 | 0
Cardiac failure acute (Cardiac disorders) | 1 | 0
Cardiac failure congestive (Cardiac disorders) | 1 | 0
Cardiogenic shock (Cardiac disorders) | 1 | 0
Ventricular arrhythmia (Cardiac disorders) | 1 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 0
Haematochezia (Gastrointestinal disorders) | 1 | 0
Large intestine perforation (Gastrointestinal disorders) | 1 | 0
Pneumatosis intestinalis (Gastrointestinal disorders) | 1 | 0
Asthenia (General disorders) | 1 | 0
Sudden cardiac death (General disorders) | 1 | 0
Cholecystitis (Hepatobiliary disorders) | 1 | 0
Ischaemic hepatitis (Hepatobiliary disorders) | 1 | 0
COVID-19 (Infections and infestations) | 2 | 0
Clostridium difficile infection (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 1 | 0
Alcohol poisoning (Injury, poisoning and procedural complications) | 0 | 1
Fall (Injury, poisoning and procedural complications) | 1 | 0
Ejection fraction decreased (Investigations) | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 0
Hormone receptor positive breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Dyskinesia (Nervous system disorders) | 1 | 0
Embolic stroke (Nervous system disorders) | 1 | 0
Syncope (Nervous system disorders) | 2 | 0
Device inappropriate shock delivery (Product Issues) | 1 | 0
Device lead damage (Product Issues) | 1 | 0
Mental status changes (Psychiatric disorders) | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 1 | 0
Nephrolithiasis (Renal and urinary disorders) | 1 | 0
Ureterolithiasis (Renal and urinary disorders) | 1 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hypovolaemic shock (Vascular disorders) | 1 | 0
Peripheral venous disease (Vascular disorders) | 1 | 0
Shock haemorrhagic (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Mavacamten (N=108) | Placebo (N=55)
Atrial fibrillation (Cardiac disorders) | 13 | 0
Palpitations (Cardiac disorders) | 14 | 2
Ventricular tachycardia (Cardiac disorders) | 1 | 5
Constipation (Gastrointestinal disorders) | 9 | 2
Diarrhoea (Gastrointestinal disorders) | 7 | 2
Nausea (Gastrointestinal disorders) | 9 | 1
Chest discomfort (General disorders) | 6 | 2
Chest pain (General disorders) | 7 | 1
Fatigue (General disorders) | 18 | 2
Bronchitis (Infections and infestations) | 7 | 1
COVID-19 (Infections and infestations) | 39 | 2
Upper respiratory tract infection (Infections and infestations) | 15 | 0
Urinary tract infection (Infections and infestations) | 15 | 1
Ejection fraction decreased (Investigations) | 12 | 0
SARS-CoV-2 test positive (Investigations) | 9 | 1
Gout (Metabolism and nutrition disorders) | 6 | 0
Hyperlipidaemia (Metabolism and nutrition disorders) | 6 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 13 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 6 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 6 | 1
Dizziness (Nervous system disorders) | 16 | 3
Headache (Nervous system disorders) | 11 | 5
Syncope (Nervous system disorders) | 6 | 0
Anxiety (Psychiatric disorders) | 8 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 7 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 11 | 3
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 10 | 2
Rash (Skin and subcutaneous tissue disorders) | 7 | 0
Hypertension (Vascular disorders) | 10 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing, but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-06-30): https://cdn.clinicaltrials.gov/large-docs/72/NCT04349072/Prot_SAP_000.pdf